CLINICAL TRIAL: NCT03168373
Title: Effect of Intensive Language Therapy in Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, MD, PhD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-07-147
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Rehabilitation; Language
MeSH Terms: conditions — Stroke; Language

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive group (Experimental): language rehabilitation therapy by language therapist for 1 hours on every working day for 4 weeks
  Interventions: Procedure: language rehabilitation therapy
- Conventional group (Active Comparator): language rehabilitation therapy by language therapist for 30 minutes on every working day for 4 weeks
  Interventions: Procedure: language rehabilitation therapy

INTERVENTIONS:
Procedure: language rehabilitation therapy — language therapy is language rehabilitation by language therapist during subacute phase in stroke patients

SUMMARY:
Early stroke rehabilitation is known to be an effective and essential therapy in gaining functional independence and preventing complications. However, there was no consensus of proper amount of language rehabilitation in stroke patients. In this study, the investigators investigated the effects of the intensive language rehabilitation during subacute phase to improve language function in patients with first-ever strokes.

DETAILED DESCRIPTION:
Intensive language rehabilitation group - language rehabilitation therapy by language therapist for 1 hours on every working day for 4 weeks

Conventional language rehabilitation group

- language rehabilitation therapy by language therapist for 30 minutes on every working day for 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Acute first-ever stroke
* Left hemispheric stroke
* Korean version of Frenchay Aphasia Screening Test(K-FAST) < 25 (less than 65 years old), K-FAST <20 (65 years old and more than 65 years old) at 7 days after stroke onset
* Right handedness

Exclusion Criteria:

* Transient ischemic stroke

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Korean version-Western Aphasia Battery (AQ) | Change of Korean version- Western Aphasia Battery after language rehabilitation for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang WH, Sohn MK, Lee J, Kim DY, Lee SG, Shin YI, Oh GJ, Lee YS, Joo MC, Han EY, Kim YH. Korean Stroke Cohort for functioning and rehabilitation (KOSCO): study rationale and protocol of a multi-centre prospective cohort study. BMC Neurol. 2015 Mar 25;15:42. doi: 10.1186/s12883-015-0293-5. PMID 25886039